CLINICAL TRIAL: NCT07193407
Title: Feasibility and Safety Study to Evaluate the Sensing and Stimulation Performance of a Personalised Sacral Neuromodulation (SNM) System for Refractory Overactive Bladder
Brief Title: INOPASE - Performance and Safety Study of a Personalised SNM System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: INOPASE Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PoC-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INOPASE Sacral Neuromodulation System 01 (INO-SNM-01) (Experimental): Participants are implanted with the Trial Lead and undergo 2 days of monitoring in hospital with the INO-SNM-01 System.
  Interventions: Device: Sacral Neuromodulation System

INTERVENTIONS:
Device: Sacral Neuromodulation System — INOPASE Sacral Neuromodulation System (INO-SNM-01) for treatment of overactive bladder.

SUMMARY:
The goal of this clinical trial is to learn whether a new sacral neuromodulation (SNM) system (INO-SNM-01) can safely and effectively sense bladder nerve activity and provide stimulation to help manage symptoms of refractory overactive bladder in adult women aged 18-70 who have not responded to standard treatments.

The main questions it aims to answer are:

* Is there a clear relationship between bladder nerve activity and patient-reported urgency sensations?
* Can targeted stimulation based on bladder nerve activity reduce overactive bladder symptoms?
* Is the INO-SNM-01 System safe to use?

Researchers will not use a comparison group in this study. Instead, all participants will receive the investigational device to see if it works as intended.

Participants will undergo surgery to have a temporary trial lead implanted near the sacral nerve and spend up to 2 days in hospital for monitoring and testing to assess the device sensing and stimulation capabilities.

Up to 10 participants will take part in this first-in-human feasibility study at a single site in Australia.

ELIGIBILITY:
Inclusion Criteria:

* Adult female participants between 18 and 70 years of age
* Diagnosed with refractory overactive bladder that is resistant to behavioural therapy and/or pharmacotherapy, for at least 12 weeks
* Experience at least 3 urgency episodes within a 24-hour period from the past 3 consecutive days (reported in a bladder diary)
* Baseline of greater than 7 on the Overactive Bladder Symptom Score (OABSS)
* Baseline score of greater than 12 on the International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS)
* Willing to receive SNM therapy
* Willing to provide free and Informed consent to participate in the clinical investigation
* Able to understand all study instructions, willing to attend all study visits, and likely to comply with all study procedures

Exclusion Criteria:

* Participants who are diagnosed with stress urinary incontinence
* Received tibial nerve stimulation therapy within the past 3 months
* Received treatment of urinary symptoms with botulinum toxin in the past 9 months or any plan to have botulinum toxin treatment during the study
* Have neurological conditions such as dementia, multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury
* Participants who presently have, or are at high risk of urinary tract infection
* Have uncontrolled systemic disease or comorbidities which may affect bladder function (for example diabetes, hypertension, cancer)
* Implanted with a neurostimulator, pacemaker, or defibrillator
* Participation in another interventional drug or device clinical trial concurrently or concluding within 30 days of screening
* Women who are pregnant
* Participants with known history of allergies to materials in contact with tissue for this study (i.e. adhesive dressing patch, silicone)
* Have implanted devices that contain metallic components
* Any other clinical or social reason that, in the opinion of the investigator could restrict a participant's ability to successfully meet the study objectives

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Correlation between bladder afferent nerve activity measured by the INO-SNM-01 and patient reported urgency sensation (Feeling Indicator measure) | From device implantation to the end of treatment 2 days
  Success is defined as the ability of the INO-SNM-01 device to detect an increase in nerve activity (mV) as measured by the INO-SNM-01 when the participant reports 'Urgency' on the wireless input Feeling Indicator device.
  The Feeling Indicator allows patients to record their urgency sensations as 'Desire to urinate', 'Loss of desire to urinate', 'Urgency' or 'Urination' in real-time throughout the test period.

SECONDARY OUTCOMES:
Evaluation of whether timely stimulation by the INO-SNM-01 device correlates with 'Loss of desire to urinate' as measured by the Feeling Indicator | From device implantation to the end of treatment 2 days
  The Feeling Indicator device allows patients to record their urgency sensations as 'Desire to urinate', 'Loss of desire to urinate', 'Urgency' or 'Urination' in real-time throughout the test period.
Evaluation of whether timely stimulation by the INO-SNM-01 device shows a reduction in bladder afferent nerve activity response when providing stimulation compared to no stimulation | From device implantation to the end of treatment 2 days
Evaluation of whether timely stimulation by the INO-SNM-01 shows a reduction in bladder pressure (cm H2O) measured by a urodynamics monitor | From device implantation to the end of treatment 2 days
Evaluation of whether timely stimulation by the INO-SNM-01 device shows an increase in urinary volume (mL) during each urination cycle as measure by a urodynamics monitor. | From device implantation to the end of treatment 2 days
Evaluation of whether timely stimulation using the INO-SNM-01 device shows an increase in time between urination cycles (minutes) as reported by the Feeling Indicator | From device implantation to the end of treatment 2 days
  Time of urination is recorded when the participant reports the 'Urination' state on the Feeling Indicator during testing.
  Time between urination cycles is calculated as the difference between 2 consecutive urination times.
Incidence of Adverse Events | From device implantation to the end of treatment 2 days
  Evaluation of device safety profile through adverse event reporting during device implantation, testing or explantation.

CONTACTS AND LOCATIONS:
Overall Officials: Wiliam Lynch, Principal Investigator — St George Urology
Locations (2):
- Australia (2):
  - St George Private Hospital, Kogarah, New South Wales
  - St George Urology, Kogarah, New South Wales

IPD SHARING:
Plan to Share IPD: No
No plans to publish paper outside of initial research group.